CLINICAL TRIAL: NCT04912869
Title: A Phase IB Randomized, Placebo-Controlled Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of Crovalimab for the Management of Acute Uncomplicated Vaso-Occlusive Episodes (VOE) in Patients With Sickle Cell Disease (SCD)
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamics and Efficacy of Crovalimab for the Management of Acute Uncomplicated Vaso-Occlusive Episodes (VOE) in Participants With Sickle Cell Disease (SCD).
Acronym: CROSSWALK-a
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO42452; 2020-004840-27 (EudraCT Number)
Record Dates: First submitted 2021-06-02; First posted 2021-06-03 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Disease
Keywords: Vaso-occlusive episodes; Pain crisis
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crovalimab (Experimental): Participants will receive a single intravenous (IV) infusion of Crovalimab based on body weight.
  Interventions: Drug: Crovalimab
- Placebo (Placebo Comparator): Participants will receive a single IV infusion of matching Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Crovalimab — Crovalimab will be administered as a single dose of 1000 milligrams (mg) IV (for participants with a body weight between 40 kilograms (kg) and 100 kg) or 1500 mg IV (for participants with a body weight >=100 kg).
  Arms: Crovalimab
Drug: Placebo — Placebo will be administered as a single IV infusion, with an equal volume and over the same duration as weight- based crovalimab
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate crovalimab for the treatment of a sickle cell pain crisis (also known as a VOE) that requires hospitalisation in adult and adolescent participants with SCD. The primary objective of this study is safety and will additionally evaluate pharmacokinetics (how crovalimab is processed by your body), pharmacodynamics (how your body reacts to crovalimab) and the preliminary efficacy of crovalimab compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >=40 kg.
* Confirmed diagnosis of HbSS (SCD genotype of sickle cell anemia) or HbSβ0 (SCD genotype of sickle cell beta zero thalassemia).
* Vaccination against Neisseria Meningitidis serotypes A, C, W, and Y.
* Vaccinations against H. influenzae type B and S. pneumoniae.
* Participants vaccinated against SARS-CoV-2 are eligible, as long as it has been 3 days or more after inoculation with the vaccine.
* Diagnosis of an acute uncomplicated VOE, that requires admission to a hospital/acute medical facility and treatment with parenteral opioid analgesics.
* Adequate hepatic and renal function.
* Hemoglobin >=5 grams/deciliter (g/dL)
* Platelet count >=100,000/microliter (µL)
* Participants receiving SCD-directed therapies must be on a stable dose for >=28 days.
* For female participants of childbearing potential, an agreement to remain abstinent or use contraception for 322 days (approximately 10.5 months) after the dose of study treatment.

Exclusion Criteria:

* More than 10 VOEs within the last 12 months prior to presentation, that have required a medical facility visit.
* Pain related to the current VOE ongoing for >36 hours.
* Acute pain related to avascular necrosis, hepatic or splenic sequestration, or priapism.
* Pain atypical of an acute uncomplicated VOE.
* Evidence of or suspicion of ACS.
* Evidence or high suspicion of a severe systemic infection.
* Major surgery and/or hospitalization for any reason within 30 days.
* History of Neisseria meningitidis infection within 6 months prior.
* Known HIV infection with a documented CD4 count <200 cells/µL.
* Transfusion or receipt of blood products within 3 months or current participation in a chronic transfusion protocol.
* Immunized with a live attenuated vaccine within 30 days.
* History of hematopoietic stem cell transplant.
* Known or suspected hereditary complement deficiency.
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 322 days (approximately 10.5 months) after the study drug administration.
* Participation in another interventional treatment study with an investigational agent or use of any experimental therapy within the prior 28 days or within five half-lives of that investigational product, whichever was greater.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-26 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Baseline up to Day 84
Percentage of Participants with Infusion-Related Reactions and Hypersensitivity | Baseline up to Day 84

SECONDARY OUTCOMES:
Time to Improvement of the Primary Acute Uncomplicated VOE From Baseline | Baseline up to Day 84
Total Cumulative Opioid Dose From Baseline | Baseline up to Day 84
Time to Discontinuation of all Parenteral Opioids From Baseline | Baseline up to Day 84
Time to Readiness For Hospital Discharge From Baseline | Baseline up to Day 84
Time to Hospital Discharge From Baseline | Baseline up to Day 84
Time to a Confirmed Decrease in Pain Score of at Least 2 Points From the Maximal Pre-dose Pain Score | Baseline up to Day 84
Change in Pain Score From the Maximal Pre-dose Pain Score to the Score at Hospital Discharge | Baseline up to Day 84
Percentage of Participants who Develop Acute Chest Syndrome (ACS) | Baseline up to Day 28
Percentage of Participants Requiring Intensive Care Unit (ICU)/Critical Care Admission for SCD-related Complications | Baseline up to Day 84
Percentage of Participants Requiring Blood Transfusion for SCD-related Complications | Baseline up to Day 84
Readmission Rate for a VOE or VOE-related Event Within 28 days of Discharge of the Primary Acute Uncomplicated VOE | Baseline up to Day 84
Serum Concentrations of Crovalimab Over Time | Baseline up to Day 84
Change in PD Biomarkers Including Complement Activity (CH50) Over Time | Baseline up to Day 84
  Assessed by a Liposome Immunoassay (LIA)
Change Over Time in Free C5 Concentration | Baseline up to Day 84
Change Over Time in Soluble Complement 5b 9 (sC5b-9) Concentration | Baseline up to Day 84
Percentage of Participants with Anti-Drug Antibodies to Crovalimab | Baseline up to Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- United States (2):
  - Children'S Healthcare of Atlanta, Atlanta, Georgia
  - Icahn School of Medicine at Mount Sinai, New York, New York
- Brazil (2):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
- CHU Henri Mondor, Créteil, France
- Azienda Ospedaliera di Verona-Policlinico G.B. Rossi, Verona, Veneto, Italy
- Kenya (2):
  - International Cancer Institute (ICI), Eldoret
  - Gertrude's Children Hospital, Nairobi
- Lebanon (2):
  - American University of Beirut - Medical Center, Beirut
  - Hopital Nini, Tripoli
- Amsterdam UMC Location VUMC, Amsterdam, Netherlands
- Charlotte Maxeke Johannesburg Hospital, Johannesburg, South Africa
- Spain (3):
  - Hospital General Univ. Gregorio Maranon, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).